CLINICAL TRIAL: NCT07199140
Title: The Effect of Haptonomy Practice on Body Functionality Appreciation and Childbirth Self-Efficacy in Pregnant Women
Acronym: HAP-Func-Eff
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nazlı BALTACI, Associate Professor, phD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GaziosmanpasaU-MUDUT-001; 2025090597 (Other: Ondokuz Mayıs University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-08; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pregnant Women
Keywords: Haptonomy; Pregnancy; Body functionality appreciation; Vaginal birth; Prenatal care; Birth self-efficacy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled, parallel-group interventional study designed to evaluate the effects of haptonomy on pregnant women's body functionality appreciation and childbirth self-efficacy. Participants in the intervention group will receive four haptonomy sessions, while the control group will receive standard prenatal care. Pre- and post-intervention assessments will be conducted to measure outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: No other parties beyond those listed above are blinded in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haptonomy Intervention (Experimental): Participants receive four sessions of haptonomy during pregnancy.
  Interventions: Behavioral: Haptonomy
- Control (No Intervention): Participants receive routine prenatal care without additional intervention

INTERVENTIONS:
Behavioral: Haptonomy — Pregnant participants will receive a four-session haptonomy intervention, each lasting approximately 45 minutes. The sessions aim to enhance body awareness, reduce childbirth-related anxiety, and support birth self-efficacy. The intervention includes breathing exercises, relaxation techniques, and activities promoting maternal-fetal interaction.
  Arms: Haptonomy Intervention

SUMMARY:
Study Type and Aim:

This clinical study aims to examine the effects of haptonomy practices on appreciation of bodily functionality and childbirth self-efficacy among healthy pregnant women. The study seeks to determine whether haptonomy can enhance these two outcomes.

Key Research Questions:

Do haptonomy practices increase appreciation of bodily functionality in pregnant women? Do haptonomy practices increase childbirth self-efficacy in pregnant women?

Comparison:

Researchers will compare an intervention group receiving haptonomy sessions with a control group receiving only routine prenatal care to evaluate the effects of the intervention.

Participants will:

Participants will provide written informed consent to take part in the study. Pregnant women in the intervention group will attend four haptonomy sessions, each lasting approximately 45 minutes and held at 7-day intervals. Sessions will include practices to enhance body awareness, relaxation techniques, connecting with the baby, and affirmations supporting bodily functionality and childbirth self-efficacy.

Pregnant women in the control group will receive routine prenatal care and follow-up only.

All participants will complete pretest and posttest measures assessing appreciation of bodily functionality and childbirth self-efficacy.

Keywords: Haptonomy, Vaginal birth, Pregnancy, Prenatal care, Body functionality appreciation, Birth self-efficacy

DETAILED DESCRIPTION:
Introduction:

Despite the World Health Organization's recommendation that cesarean section rates should ideally be between 10-15%, this limit has already been exceeded in many countries. Globally, cesarean birth rates have increased significantly over the last few decades. While the overall cesarean rate was around 5-7% in the 1980s, it had risen to 21-23% by the 2000s. In countries such as Turkey, cesarean rates exceed 60%, ranking among the highest worldwide.

The rise in cesarean rates is influenced by factors such as fear of childbirth, desire for control, wish for a positive birth experience, negative past birth experiences, media portrayals, and healthcare professionals' guidance. Additionally, the weakening of the belief that childbirth is a "physiological process," perceiving it instead as a medical event, women's distancing from body knowledge and birth experience, and their being placed in a passive role during childbirth are also reasons for preferring cesarean delivery.

Cesarean delivery, when chosen beyond medical necessity, creates short- and long-term risks for maternal and infant health. Therefore, healthcare professionals and society should acknowledge that normal birth is safe and natural, and conduct awareness and education programs. Nurses are responsible for reducing prenatal anxiety and fears, as well as providing communication and supportive techniques during childbirth. It is known that non-pharmacological methods applied by nurses reduce labor pain and anxiety, shorten the process, and increase rates of normal birth. Thus, nurses' accurate guidance and awareness practices during pregnancy and childbirth are of critical importance.

One of the practices that supports expectant mothers during pregnancy and beyond is haptonomy, which enhances confidence in the body by fostering emotional connection through touch throughout pregnancy. This approach enables women to better perceive their bodies, adapt to bodily changes, and develop positive awareness of their vital functions. Haptonomy contributes to women feeling secure and supported through bodily sensations, strengthens psychological resilience, and reduces fears and anxieties about normal birth. It also allows women to express their thoughts, needs, and emotions related to pregnancy and childbirth.

During pregnancy, the female body is highlighted through complex functions such as fertility and childbirth. A positive attitude toward the body during this period includes respect for fertility, growth, and birth functions. This approach supports body acceptance and the development of positive body image, thereby increasing body satisfaction. Moreover, it strengthens resilience by enhancing the ability to cope with difficulties. Women with high body satisfaction experience less fear and anxiety regarding normal childbirth and report more positive birth experiences.

Confidence in one's body fosters greater belief in one's abilities and increases self-efficacy. Self-efficacy enhances performance, resilience, and motivation. In the context of pregnancy, a woman's positive attitude toward her body can positively affect overall health, psychological well-being, and the experience of normal childbirth. Therefore, haptonomy is considered to enhance appreciation of bodily functionality, respect for the body, and self-efficacy regarding childbirth.

In recent years, studies investigating the use and effects of haptonomy during pregnancy have increased worldwide. Haptonomy has been shown to improve prenatal parental attachment, adjustment to pregnancy, and acceptance of pregnancy, while reducing stress, anxiety, and fear of childbirth. However, there are no studies examining the effects of haptonomy on appreciation of bodily functionality and childbirth self-efficacy.

Aim of the Study:

To examine the effects of haptonomy practices on appreciation of bodily functionality and childbirth self-efficacy among pregnant women.

Hypotheses:

H0: Haptonomy practices for pregnant women do not have a significant effect on levels of appreciation of bodily functionality and childbirth self-efficacy.

H11: Haptonomy practices for pregnant women significantly increase appreciation of bodily functionality.

H12: Haptonomy practices for pregnant women significantly increase childbirth self-efficacy.

Method:

Type of Study:

This research is a randomized controlled experimental study designed with a single-blind, parallel, pretest-posttest control group design.

Population and Sample The study population consists of healthy pregnant women who apply to the obstetrics outpatient clinic of Tokat/Erbaa State Hospital. The sample will include 80 healthy pregnant women who meet the research criteria and volunteer to participate. Sample size was determined by power analysis using the G-Power 3.1.9.7 program. According to the analysis, 72 participants were required, with 36 in each group. Considering at least 10% possible data loss, 40 participants were included in each of the intervention and control groups.

Randomization and Blinding:

Women who meet the inclusion criteria will be randomly assigned to intervention and control groups according to a list generated by simple randomization. The randomization list will be created by computer software, and assignments will be carried out by a statistics specialist. Participants will not know which group they belong to. In addition, groups will be coded when transferring data into SPSS software to ensure statistical blinding. To prevent interaction among participants, pregnant women will be admitted individually to the outpatient clinic, and interventions will be conducted in the prenatal education unit without communication with other pregnant women.

Procedure:

Pilot Study:

A pilot study will be conducted with 8 women (10% of the sample). After the pilot, the comprehensibility, adequacy, and applicability of the data collection form and procedure will be evaluated, and necessary adjustments will be made. Women participating in the pilot will not be included in the main study.

Data Collection:

After being informed about the study, eligible pregnant women who volunteer will provide written consent. They will then be randomly assigned to one of the two groups. All participants will first complete a personal information form, and levels of appreciation of bodily functionality and childbirth self-efficacy will be assessed before (pretest) and after (posttest) the intervention. Data will be collected face-to-face by the researcher based on participants' self-reports. Routine care, treatment, and follow-up will not be interrupted during the research.

Intervention Group:

Pregnant women in the intervention group will receive haptonomy practices in four sessions, each lasting approximately 45 minutes, held at 7-day intervals. Sessions will be conducted by the researcher, who has received special training in haptonomy. The training content will include practices to enhance body awareness, relaxation techniques, connecting with the baby, and affirmations aimed at strengthening bodily functionality and self-efficacy in childbirth. The goal is to reinforce women's relationship with their bodies, promote positive perceptions of childbirth, and support belief in their ability to actively manage the birthing process.

Control Group:

Pregnant women in the control group will receive only routine prenatal care and follow-up. As part of the hospital's routine prenatal monitoring, maternal history will be obtained, necessary tests and examinations will be conducted, and maternal-fetal well-being will be assessed.

Statistical Analysis:

Data will be analyzed using IBM SPSS Statistics 21.0. Descriptive statistics will include frequency, percentage, mean, standard deviation, median, minimum, and maximum values. Normality of distribution will be evaluated using the Shapiro-Wilk test and skewness-kurtosis values. For normally distributed data, independent samples t-test and paired samples t-test will be used; for non-normally distributed data, Mann-Whitney U test and Wilcoxon signed-rank test will be applied. Statistical significance will be set at p < 0.05.

Ethical Considerations:

This research will be conducted in accordance with ethical principles after receiving approval from the Clinical Research Ethics Committee of Ondokuz Mayıs University and obtaining necessary institutional permissions. Written informed consent will be obtained from women who volunteer to participate. Permissions for the use of study scales have been secured. The research protocol has been prepared in line with the SPIRIT guidelines, and reporting will follow the CONSORT checklist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Spontaneous pregnancy at 28 weeks of gestation
* Primiparous (first pregnancy)
* Able to read and write in Turkish
* Healthy singleton pregnancy

Exclusion Criteria:

* Any health problems in the mother or fetus
* History of complications during pregnancy
* Diagnosed psychiatric disorders or use of psychiatric medication
* Any physical, mental, or cognitive disabilities

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The sociodemographic characteristics of the participants and their homogeneous distribution according to the experimental and control groups | baseline
  Pregnancy Introductory Form: The pregnancy introductory form, developed based on the literature, was designed to evaluate the demographic and obstetric characteristics of individuals during pregnancy, their birth preferences, fears, social support status, and similar factors. The form consists of a total of 15 questions.
Body Functionality Appreciation Scale: | 12 weeks
  This unidimensional 7-item scale measures individuals' appreciation of their body's functionality. It evaluates psychological aspects such as body functionality awareness, body positivity, and body acceptance. The scale is scored on a 5-point Likert scale (1=Strongly disagree, 5=Strongly agree), with total scores ranging from 7 to 35. Higher scores indicate a greater level of appreciation and respect for what one's body can do. The Turkish adaptation reported a Cronbach's alpha of 0.83.
Birth Self-Efficacy Inventory: | 12 weeks
  This inventory measures self-efficacy levels during labor. It consists of two subscales: outcome expectancy (OE) and efficacy expectancy (EE), each containing 16 items. Total scores range from 32 to 320. Responses are rated on a 1-10 Likert scale. In the OE subscale, 1 means "not at all useful" and 10 means "very useful." In the first 13 items of the EE subscale, 1 means "completely sure" and 10 means "not at all sure," while items 14-16 are scored in reverse: 1 means "not at all sure" and 10 means "completely sure." Items 1-13 of the EE subscale are reverse-scored. The overall Cronbach's alpha reliability coefficient of the inventory is 0.82.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa University, Erbaa Faculty of Health Sciences, Erbaa, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study is limited to internal analysis and participant confidentiality will be maintained.